CLINICAL TRIAL: NCT03363919
Title: Glutamatergic and GABAergic Biomarkers in rTMS for Adolescent Depression
Brief Title: Biomarkers in Repetitive Transcranial Magnetic Stimulation (rTMS) for Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Neuronetics (Other)
Responsible Party: Principal Investigator, Paul E. Croarkin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-004958; 1R01MH113700-01 (NIH)
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
Keywords: adolescent; biomarkers
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: In both phases of the study (phase I and phase II) participants and study team members completing clinical rating scales will be blinded to treatment assignment. The study team member completing clinical rating scales and analyzing TMS neurophysiology measures will not be allowed in the treatment suite during therapeutic rTMS sessions (10 Hz, 1 Hz, iTMS, or cTBS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 1 Hz left prefrontal rTMS (Active Comparator): 36 sessions of 1 Hz rTMS at 120% motor threshold applied to the left prefrontal cortex. Each session is 2400 continuous pulses.
  Interventions: Device: NeuroStar TMS Therapy® System; Device: NeuroStar XPLOR®
- 10 Hz left prefrontal rTMS (Active Comparator): 36 sessions of 10 Hz rTMS at 120% motor threshold applied to the left prefrontal cortex. Each session is 2400 pulses with 4 seconds on and 36 seconds off.
  Interventions: Device: NeuroStar TMS Therapy® System; Device: NeuroStar XPLOR®

INTERVENTIONS:
Device: NeuroStar TMS Therapy® System — The NeuroStar TMS Therapy® System is a computerized electromechanical instrument that produces and delivers brief duration, rapidly alternating (pulsed) magnetic fields to induce electrical currents in localized regions of the cerebral cortex. It is a non-invasive tool used for the treatment of Participants with Major Depressive Disorder (MDD) who have not achieved sufficient clinical benefit from antidepressant pharmacotherapy.
Device: NeuroStar XPLOR® — NeuroStar XPLOR® is a clinical research option for the NeuroStar TMS Therapy System that provides features necessary to conduct randomized controlled trials and other TMS research.

SUMMARY:
The Researchers are going to gather information regarding the use of rTMS as a treatment for depression in adolescents with Major Depressive Disorder. The researchers also hope to learn if measures of brain activity (cortical excitability and inhibition) collected with transcranial magnetic stimulation (TMS) can be used to identify which patients will benefit from certain types of rTMS treatment.

DETAILED DESCRIPTION:
Phase I is a double-blind, randomized, biomarker-stratified trial of 1 Hz vs. 10 Hz rTMS. Phase II is for participants who do not respond to Phase I treatment and is a biomarker guided, double-blind trial of continuous vs intermittent theta burst stimulation (TBS). Please note that transcranial magnetic stimulation (TMS) biomarkers will be collected in this protocol during the course of the proposed interventions. Participants in Phase I will be offered enrollment in a separate protocol with baseline and posttreatment 7 Tesla Magnetic Resonance Imaging (MRI) and Magnetic Resonance Spectroscopy (MRS) scans

ELIGIBILITY:
Inclusion Criteria:

* Depressed adolescent participants will have a primary diagnoses of MDD based on a clinical and structured interview with the MINI
* Depression symptoms severity of a 40 or greater based on evaluation with the Children's Depression Rating Scale Revised (CDRS-R) at screening and baseline visits. Further, the total score of the baseline CDRS-R score must not have had a 25% or greater decrease from the screening CDRS-R score
* The duration of the current episode of depression must be 4 weeks or more but 3 years or less.
* For any participant currently receiving antidepressant medication, the referring clinician must determine that insufficient benefit is being received from this treatment and it is clinically appropriate to discontinue the existing antidepressant.
* Participants in psychotherapy are eligible provided that this was initiated 4 weeks prior to enrollment and that the frequency of visits will be maintained during study participation.

Exclusion criteria:

* The following psychiatric comorbidities are exclusionary: psychotic disorders, bipolar disorders, anorexia nervosa, bulimia nervosa, and substance use disorders within the past year (with the exception of caffeine and tobacco)
* A positive urine drug screen at baseline
* Seizure history
* Family history of epilepsy in a first degree relative
* Head trauma with loss of consciousness for greater than 5 minutes
* Any true positive findings on the rTMS safety screening form.
* Any concurrent psychotropic medications (for potential participants receiving antidepressants or psychotropic medications, the referring clinician must determine that insufficient benefit is being received from the treatment and if clinically appropriate, discontinue existing antidepressants and other psychotropic medications)
* Prohibited concomitant medications (See Appendix A)
* Pregnancy or suspected pregnancy in female Participants (assessed with urine pregnancy test)
* Conductive, ferromagnetic, or other magnetic-sensitive metals implanted in the subject's head within 30 cm of the treatment coil excluding the mouth that cannot safely be removed. Examples include cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewelry and hair barrettes.
* Prior brain surgery
* Risk for increased intracranial pressure such as a brain tumor
* Any unstable medical condition
* History of treatment with ECT or TMS Therapy for any disorder
* Use of any investigational drug within 4 weeks of the baseline visit
* Initiation of a new psychotherapeutic treatment within the past 4 weeks
* Suicide attempt within the previous 6 months that required medical treatment or ≥ 2 attempts in the past 12 months, or has a clear cut plan for suicide and states that he/she cannot guarantee that he/she will inform a family member or call his/her psychiatrist or the investigator if the impulse to implement the plan becomes substantial during the study; or, in the investigator's opinion, is likely to attempt suicide within the next 6 months.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Croarkin, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wall CA, Croarkin PE, Maroney-Smith MJ, Haugen LM, Baruth JM, Frye MA, Sampson SM, Port JD. Magnetic Resonance Imaging-Guided, Open-Label, High-Frequency Repetitive Transcranial Magnetic Stimulation for Adolescents with Major Depressive Disorder. J Child Adolesc Psychopharmacol. 2016 Sep;26(7):582-9. doi: 10.1089/cap.2015.0217. Epub 2016 Feb 5. PMID 26849202
- [Background] Croarkin PE, Nakonezny PA, Wall CA, Murphy LL, Sampson SM, Frye MA, Port JD. Transcranial magnetic stimulation potentiates glutamatergic neurotransmission in depressed adolescents. Psychiatry Res Neuroimaging. 2016 Jan 30;247:25-33. doi: 10.1016/j.pscychresns.2015.11.005. Epub 2015 Nov 27. PMID 26651598
- [Background] Croarkin PE, Wall CA, Lee J. Applications of transcranial magnetic stimulation (TMS) in child and adolescent psychiatry. Int Rev Psychiatry. 2011 Oct;23(5):445-53. doi: 10.3109/09540261.2011.623688. PMID 22200134
- [Background] Wall CA, Croarkin PE, Sim LA, Husain MM, Janicak PG, Kozel FA, Emslie GJ, Dowd SM, Sampson SM. Adjunctive use of repetitive transcranial magnetic stimulation in depressed adolescents: a prospective, open pilot study. J Clin Psychiatry. 2011 Sep;72(9):1263-9. doi: 10.4088/JCP.11m07003. PMID 21951987
- [Background] Croarkin PE, Nakonezny PA, Husain MM, Melton T, Buyukdura JS, Kennard BD, Emslie GJ, Kozel FA, Daskalakis ZJ. Evidence for increased glutamatergic cortical facilitation in children and adolescents with major depressive disorder. JAMA Psychiatry. 2013 Mar;70(3):291-9. doi: 10.1001/2013.jamapsychiatry.24. PMID 23303429
- [Background] Donaldson AE, Gordon MS, Melvin GA, Barton DA, Fitzgerald PB. Addressing the needs of adolescents with treatment resistant depressive disorders: a systematic review of rTMS. Brain Stimul. 2014 Jan-Feb;7(1):7-12. doi: 10.1016/j.brs.2013.09.012. PMID 24527502
- [Background] Krishnan C, Santos L, Peterson MD, Ehinger M. Safety of noninvasive brain stimulation in children and adolescents. Brain Stimul. 2015 Jan-Feb;8(1):76-87. doi: 10.1016/j.brs.2014.10.012. Epub 2014 Oct 28. PMID 25499471
- [Derived] Delaney K, Nakonezny PA, Buyuktaskin D, Carrasco LS, Athreya AP, Romanowicz M, Shekunov J, Vande Voort JL, Croarkin PE. Trajectories of Irritability Improvement in Depressed Adolescents Treated With 1 Hz and 10 Hz Transcranial Magnetic Stimulation. J Clin Psychiatry. 2025 Apr 9;86(2):24m15684. doi: 10.4088/JCP.24m15684. PMID 40215375
- [Derived] Lewis CP, Nakonezny PA, Sonmez AI, Ozger C, Garzon JF, Camsari DD, Yuruk D, Romanowicz M, Shekunov J, Zaccariello MJ, Vande Voort JL, Croarkin PE. A Dose-Finding, Biomarker Validation, and Effectiveness Study of Transcranial Magnetic Stimulation for Adolescents With Depression. J Am Acad Child Adolesc Psychiatry. 2025 Oct;64(10):1179-1191. doi: 10.1016/j.jaac.2024.08.487. Epub 2024 Sep 6. PMID 39245178
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Hz Left Prefrontal rTMS: 36 sessions of 1 Hz rTMS at 120% motor threshold were applied to the left prefrontal cortex. Each session was 2400 continuous pulses.
  NeuroStar TMS Therapy® System: The NeuroStar TMS Therapy® System is a computerized electromechanical instrument that produces and delivers brief duration, rapidly alternating (pulsed) magnetic fields to induce electrical currents in localized regions of the cerebral cortex. It is a non-invasive tool used for the treatment of Participants with Major Depressive Disorder (MDD) who have not achieved sufficient clinical benefit from antidepressant pharmacotherapy.
  NeuroStar XPLOR®: NeuroStar XPLOR® is a clinical research option for the NeuroStar TMS Therapy System that provides features necessary to conduct randomized controlled trials and other TMS research.
- 10 Hz Left Prefrontal rTMS: 36 sessions of 10 Hz rTMS at 120% motor threshold were applied to the left prefrontal cortex. Each session was 2400 pulses with 4 seconds on and 36 seconds off.
  NeuroStar TMS Therapy® System: The NeuroStar TMS Therapy® System is a computerized electromechanical instrument that produces and delivers brief duration, rapidly alternating (pulsed) magnetic fields to induce electrical currents in localized regions of the cerebral cortex. It is a non-invasive tool used for the treatment of Participants with Major Depressive Disorder (MDD) who have not achieved sufficient clinical benefit from antidepressant pharmacotherapy.
  NeuroStar XPLOR®: NeuroStar XPLOR® is a clinical research option for the NeuroStar TMS Therapy System that provides features necessary to conduct randomized controlled trials and other TMS research.
Period: Overall Study
Arm/Group | 1 Hz Left Prefrontal rTMS | 10 Hz Left Prefrontal rTMS
Started | 23 | 24
Completed | 22 | 19
Not Completed | 1 | 5
Not completed — Withdrawal by subject - did not receive allocated intervention | 0 | 1
Not completed — Withdrawal by subject - discontinued intervention prior to week 1 | 1 | 4

BASELINE CHARACTERISTICS:
Population: 1 subject in the 1 Hz arm and 5 subjects in 10 hz arm were excluded in the analysis population due to subject withdrawal.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Hz Left Prefrontal rTMS | 10 Hz Left Prefrontal rTMS | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.68 (1.83) | 15.89 (1.05) | 15.78 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 20 | 16 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 17 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Total Children's Depression Rating Scale, Revised (CDRS-R) Score
Description: CDRS-R is a 17-item scale, with items ranging from 1 to 5 or 1 to 7 (possible total score from 17 to 113), rated by a clinician via interviews with the child and parent. A score of ≥40 is indicative of depression, whereas a score ≤28 is often used to define remission (minimal or no symptoms)
Time Frame: 6 weeks
Population: Data was not collected or analyzed for one subject in the 1 Hz arm and five subjects in the 10 Hz arm
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- 1 Hz Left Prefrontal rTMS: 36 sessions of 1 Hz rTMS at 120% motor threshold were applied to the left prefrontal cortex. Each session was 2400 continuous pulses.
  NeuroStar TMS Therapy® System: The NeuroStar TMS Therapy® System is a computerized electromechanical instrument that produces and delivers brief duration, rapidly alternating (pulsed) magnetic fields to induce electrical currents in localized regions of the cerebral cortex. It is a non-invasive tool used for the treatment of Participants with MDD who have not achieved sufficient clinical benefit from antidepressant pharmacotherapy.
  NeuroStar XPLOR®: NeuroStar XPLOR® is a clinical research option for the NeuroStar TMS Therapy System that provides features necessary to conduct randomized controlled trials and other TMS research.
- 10 Hz Left Prefrontal rTMS: 36 sessions of 10 Hz rTMS at 120% motor threshold were applied to the left prefrontal cortex. Each session was 2400 pulses with 4 seconds on and 36 seconds off.
  NeuroStar TMS Therapy® System: The NeuroStar TMS Therapy® System is a computerized electromechanical instrument that produces and delivers brief duration, rapidly alternating (pulsed) magnetic fields to induce electrical currents in localized regions of the cerebral cortex. It is a non-invasive tool used for the treatment of Participants with MDD who have not achieved sufficient clinical benefit from antidepressant pharmacotherapy.
  NeuroStar XPLOR®: NeuroStar XPLOR® is a clinical research option for the NeuroStar TMS Therapy System that provides features necessary to conduct randomized controlled trials and other TMS research.
Arm/Group | 1 Hz Left Prefrontal rTMS | 10 Hz Left Prefrontal rTMS
Number analyzed (Participants) | 22 | 19
score on a scale | 41.768 [40.034 to 43.503] | 44.541 [42.633 to 46.448]

2. Secondary Outcome: Change in Intracortical Facilitation (ICF)
Description: ICF measures were collected with surface electromyography. A subthreshold conditioning stimulus (CS) was set to 80% of resting motor threshold (RMT) preceding a suprathreshold test stimulus (TS), which was calibrated to produce an average motor evoked potential (MEP) of 0.5 to 1.5 millivolt peak-to-peak amplitude in the contralateral abductor pollicis brevis (APB) muscle. Conditioning stimuli were delivered to the motor cortex prior to the TS in 15 msec interstimulus intervals. Changes in TS MEP was expressed as a percentage of the mean unconditioned MEP amplitude.
Time Frame: baseline, 6 weeks
Population: Data was not collected or analyzed for one subject in the 1 Hz arm and five subjects in the 10 Hz arm
Measure: Geometric Least Squares Mean (Standard Error); unit: percentage of the mean unconditioned MEP
Arm/Group | 1 Hz Left Prefrontal rTMS | 10 Hz Left Prefrontal rTMS
Number analyzed (Participants) | 22 | 19
percentage of the mean unconditioned MEP | 1.71 (0.05) | 1.67 (0.06)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline (consent signing) to end of study for all participants, approximately 6 weeks.
Description: Adverse events were collected on all participants whether or not they received the intervention.
Arm/Group | 1 Hz Left Prefrontal rTMS | 10 Hz Left Prefrontal rTMS
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/23 | 3/24
Other Adverse Events (participants affected / at risk) | 20/23 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Hz Left Prefrontal rTMS (N=23) | 10 Hz Left Prefrontal rTMS (N=24)
blurred vision (Eye disorders) | 1 | 0
suicidal ideation (Psychiatric disorders) | 0 | 1
severe scalp pain (Nervous system disorders) | 0 | 1
left ear bleeding (Ear and labyrinth disorders) | 0 | 1
chest pain (Cardiac disorders) | 1 | 0
groin pain (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Hz Left Prefrontal rTMS (N=23) | 10 Hz Left Prefrontal rTMS (N=24)
Anxiety (Psychiatric disorders) | 0 | 1
Auditory (Ear and labyrinth disorders) | 3 | 4
Dizziness (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 11 | 12
Insomnia (Psychiatric disorders) | 3 | 2
Nausea (General disorders) | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Non-Suicidal Self injury (Psychiatric disorders) | 1 | 0
Pain or Discomfort at Treatment site (General disorders) | 12 | 15
Sedation (Nervous system disorders) | 2 | 4
Suicidal Ideation (Psychiatric disorders) | 2 | 2
Twitching during treatment (Nervous system disorders) | 1 | 5
Worsening depression (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT03363919/Prot_SAP_000.pdf